CLINICAL TRIAL: NCT00718575
Title: A Prospective, Randomized Trial to Investigate the Effects of Glucose/ Ischemic Preconditioning Donor Pre-treatment on Reperfusion Injury in Deceased-Donor Liver Transplantation
Brief Title: The Effects of Glucose/Ischemic Preconditioning on Reperfusion Injury in Deceased-Donor Liver Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: too few patients meeting current eligibility criteria
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-0587-AE
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-06

CONDITIONS: Liver Transplantation
Keywords: Liver Disease; Transplantation
MeSH Terms: conditions — Liver Diseases | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Deceased liver donors that are randomized to this arm will receive the Glucose/Ischemic Preconditioning pre-treatment intra-operatively prior to starting cold preservation of the organ
  Interventions: Procedure: Glucose/Ischemic Preconditioning Pre-treatment
- 2 (No Intervention): Neither donors nor recipients receive any intervention. All procedures will be performed according to our institution's standard of care.

INTERVENTIONS:
Procedure: Glucose/Ischemic Preconditioning Pre-treatment — A 20% dextrose+insulin infusion is administered to the liver via the mesenteric vein beginning after cannulation of the mesenteric vein and ending immediately prior to flushing with cold preservation fluid. Also, after completion of the visceral dissection but prior to cross-clamping, ischemic precondition will occur. This involves occluding the portal vein and hepatic artery to stop blood flow for 10 minutes, then restoring blood flow for 10 minutes.
  Arms: 1

SUMMARY:
Standard liver retrieval procedures for transplantation from a deceased donor inevitably result in a "reperfusion injury" to the liver tissue. The purpose of this research study is to find out whether treatment of the liver with a "preconditioning" protocol before its removal from the donor will help reduce any of this injury.

The "preconditioning" treatment being tested has two components. Firstly, a solution of glucose+insulin is infused and secondly, blood flow to the liver is stopped briefly (10 minutes) and then resumed. Both strategies, individually, have been shown to reduce liver tissue injury in human studies.

We hypothesize that combining both strategies will have a clinical benefit to patients and will improve liver function following transplant.

DETAILED DESCRIPTION:
Liver transplantation is the only chance of cure for patients with end-stage liver disease. Unfortunately, standard organ preservation results in an ischemic-reperfusion injury (IRI) at the time of graft implantation. Novel strategies have been proposed to decrease reperfusion injury and improve graft function. This study will be the first to combine both strategies in a randomized, prospective trial. The intervention will occur during the retrieval surgery prior to cold preservation. Briefly, a glucose and insulin solution will be infused via the mesenteric vein at a controlled rate. Immediately prior to cross-clamping, blood supply to the liver will be restricted for 10 minutes and then resumed for 10 minutes before beginning cold preservation. All remaining surgical procedures, including the recipient surgery, will be performed by standard techniques. The liver recipient does not directly receive any intervention during this study.

ELIGIBILITY:
Inclusion Criteria:

* Recipient 18 years of age or older
* Recipient with chronic end-stage liver disease
* Deceased donor liver transplant
* Recipient capable of providing written informed consent
* Whole organ graft from donors aged 60 years or older

Exclusion Criteria:

* Fulminant liver failure
* Objection by any other member of the retrieval team
* Split-liver grafts
* Donor that has received total parenteral nutrition within 24hr of organ retrieval Donors from whom the pancreas and/or small bowel are also being retrieved

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reperfusion injury determined by peak AST | first 24 hours post-operative

SECONDARY OUTCOMES:
Biliary Complications, infection and rejection | first month post-transplantation
graft and patient survival; length of hospital stay; length of ICU stay | 30 days and 90 days post-transplantation
Liver ATP and glycogen content; blood cytokine levels; liver gene expression of pro- and anti-apoptotic genes | immediately pre-removal and post- transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Selzner, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network (Toronto General Hospital), Toronto, Ontario, Canada